CLINICAL TRIAL: NCT04935788
Title: The Acute Postprandial Response of Blood Amino Acids in Older Adults After Consumption of Dairy Protein, Plant Protein and Their Blend
Brief Title: Postprandial Amino Acid Response After Protein Consumption
Acronym: PAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wageningen University (Other)
Collaborators: NIZO Food Research (Other); Ingredia S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NL78067.028.21
Record Dates: First submitted 2021-06-11; First posted 2021-06-23 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Milk Proteins; Pea Proteins

STUDY DESIGN:
Intervention Model Description: a randomized, single-blinded within-subject (cross-over) trial in which a group of 12 subjects receive 4 different conditions
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- milk protein (Experimental): milk protein supplement
  Interventions: Dietary Supplement: milk protein
- micellar casein (Experimental): casein supplement
  Interventions: Dietary Supplement: micellar casein
- pea protein (Experimental): pea protein supplement
  Interventions: Dietary Supplement: pea protein
- milk/pea protein (Experimental): a blend of milk and pea protein
  Interventions: Dietary Supplement: milk/pea protein blend

INTERVENTIONS:
Dietary Supplement: milk protein — milk protein supplement
  Arms: milk protein
Dietary Supplement: micellar casein — micellar casein supplement
  Arms: micellar casein
Dietary Supplement: pea protein — pea protein supplement
  Arms: pea protein
Dietary Supplement: milk/pea protein blend — milk/pea protein supplement
  Arms: milk/pea protein

SUMMARY:
Increasing muscle protein synthesis via protein-based nutrition, with or without exercise, maintains a strong, healthy muscle mass, which in turn leads to improved health, independence and functionality in older adults. There is increased interest in plant-based proteins, but these have in general a lower anabolic effect than animal proteins. Various strategies have been suggested to augment the anabolic properties of plant proteins, including using plant-animal protein blends. However, only little is known yet about the anabolic properties of such an approach. As the peripheral metabolic availability of proteins is an important aspect that has to be taken into account when screening the anabolic properties of protein sources/blends, it is the aim of this study to investigate the postprandial AA response of milk protein, micellar casein, pea protein, and a milk protein-pea protein blend in healthy older adults.

DETAILED DESCRIPTION:
Objective:

The primary objective is to quantify the postprandial area under the curve (iAUC), the maximal level (Cmax) and the time profile (Tmax) of blood amino acids after ingestion of milk protein, micellar casein, pea protein, and a milk protein-pea protein blend in healthy older adults.

Secondary objectives are to quantify the postprandial insulin response, and to quantify the potential muscular response, using an in vitro muscle cell assay, of postprandial blood derived from healthy older adults after ingestion of milk protein, micellar casein, pea protein, and a milk protein-pea protein blend.

Study design: The study is designed as a randomized, single-blinded within-subject (cross-over) trial in which a group of 12 subjects receive 4 different protein drinks.

Study population: Healthy older adults (60-80 years) Intervention (if applicable): Four different protein drinks will be investigated: milk protein, micellar casein, pea protein, and a milk protein/ pea protein blend. All drinks will contain a 20 gram protein load. All protein supplements will be mixed with 250 mL water and contain some additional non-caloric flavorings.

Main study parameters/endpoints: Postprandial blood amino acid response, up to 5 hours after consumption of a protein drink measured (incremental area under curve, Cmax and Tmax).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥60 and ≤80
* BMI ≥20 and ≤32 kg/m2
* Non-smoking
* Healthy as assessed by a lifestyle and health questionnaire ("Verklaring leefgewoonten en gezondheid") and according to the judgment of the study physician.
* Regular and normal Dutch eating habits as assessed by a lifestyle and health questionnaire (3 main meals per day)
* Veins suitable for cannulation (blood sampling)
* Voluntary participation
* Having given written informed consent
* Willing to comply with study procedures
* Accept use of all encoded data, including publication, and the confidential use and storage of all data for 15 years.
* Accept disclosure of the financial benefit of participation in the study to the authorities concerned

Exclusion Criteria:

* Participation in any clinical trial including blood sampling and/or administration of substances up to 30 days before day 1 of this study
* Having a history of medical or surgical events that may significantly affect the study outcome, including: Inflammatory bowel disease, hepatitis, pancreatitis, ulcers, gastrointestinal or rectal bleeding; major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection; known or suspected gastrointestinal disorders, colon or GI tract cancer
* Use of the following medication: glucose lowering drugs, insulin; medication that may impact gastric emptying (e.g. gastric acid inhibitors or laxatives)
* Diagnosed with diabetes, being treated for high blood glucose or increased fasting blood glucose (> 7 mmol/l in finger prick blood) as assessed during screening visit
* For men: Hb <8,5 mmol/l as assessed during screening visit; for women: Hb <7,5 mmol/l
* Use of protein supplements
* Mental status that is incompatible with the proper conduct of the study
* A self-reported reported food allergy or sensitivity to dairy or plant ingredients
* Alcohol consumption for men > 28 units/week and >4/day; for women: >21 units/week and >3/day
* Reported unexpected weight loss or weight gain of > 3 kg in the month prior to pre-study screening, or intention to lose weight during the study period
* Reported slimming or medically prescribed diet
* Recent blood donation (<1 month prior to Day 01 of the study)
* Not willing to give up blood donation during the study
* Not having a general practitioner
* Not willing to accept information-transfer concerning participation in the study, or information regarding his or her health, like laboratory results and eventual adverse events to and from his general practitioner

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
plasma AA | 5 hours
  postprandial plasma AA response

SECONDARY OUTCOMES:
Insulin | 3 hours
  postprandial insulin response

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Human Nutrition, Wageningen University, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided